CLINICAL TRIAL: NCT06059222
Title: The Optimised Use of Romozosumab Study
Acronym: OPTIMIST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-2023-505940-20-00
Record Dates: First submitted 2023-09-08; First posted 2023-09-28 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — romosozumab; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - ROMO 12 months, ZOL 12 months (Active Comparator): 90 patients 12 months of romosozumab (ROMO) followed by 12 months of zoledronate (ZOL)
  Interventions: Drug: Romosozumab; Drug: Zoledronate
- Group 2 - ROMO 6 months, ZOL 12 months, ROMO 6 months (Active Comparator): 90 patients 6 months of romosozumab followed by 12 months of zoledronate and lastly 6 months of romosozumab.
  Interventions: Drug: Romosozumab; Drug: Zoledronate
- Group 3 - ROMO 6 months, ZOL 18 months (Active Comparator): 90 patients 6 months of romosozumab followed by 18 months of zoledronate
  .
  Interventions: Drug: Romosozumab; Drug: Zoledronate

INTERVENTIONS:
Drug: Romosozumab — Romosozumab 210 mg/2.34 ml from baseline to month 11
  Other Names: Evenity
  Arms: Group 1 - ROMO 12 months, ZOL 12 months
Drug: Zoledronate — 5 mg/100 ml at month 12
  Arms: Group 1 - ROMO 12 months, ZOL 12 months
Drug: Romosozumab — 210 mg/2.34 ml from baseline to month 5 and from month 18 to month 23
  Other Names: Evenity
  Arms: Group 2 - ROMO 6 months, ZOL 12 months, ROMO 6 months
Drug: Zoledronate — 5 mg/100 ml at month 6
  Arms: Group 2 - ROMO 6 months, ZOL 12 months, ROMO 6 months
Drug: Romosozumab — 210 mg/2.34 ml from baseline to month 5
  Other Names: Evenity
  Arms: Group 3 - ROMO 6 months, ZOL 18 months
Drug: Zoledronate — 5 mg/100 ml at month 5 and month 18
  Arms: Group 3 - ROMO 6 months, ZOL 18 months

SUMMARY:
OPTIMIST is a two-year, randomised, active controlled, open-label, multicentre intervention trial. OPTIMIST includes 3 treatment groups each comprising combinations of romosozumab (ROMO) and zoledronate (ZOL) treatment used in standard doses (210 mg monthly (sc) and 5 mg yearly (iv), respectively).

The study will investigate if it is possible to maximize the effect of romosozumab by giving it in 2 periods of 6 months interrupted by zoledronate for 12 months compared to romosozumab for 12 months uninterrupted followed by zoledronate for 12 months. The investigators will also evaluate if 6 months of romosozumab followed by 18 months of zoledronate is non-inferior to the standard regimen of romosozumab for 12 months followed by zoledronate for 12 months.

DETAILED DESCRIPTION:
Recent clinical trials have demonstrated the benefit of bone anabolic treatment over no treatment or antiresorptive treatment in terms of increasing bone mineral density (BMD) and reducing fracture risk for patients with osteoporosis. However, the bone anabolic treatment is expensive and therefore restricted to a limited group of patients.

This study is based on the hypothesis that treatment with romosozumab for 6 months, zoledronate for 12 months, and romosozumab for 6 months results in larger gains in bone mineral density than treatment regimens based on romosozumab treatment for 6 or 12 months followed by zoledronate for a total of 24 months of treatment due to reappearance of the bone anabolic effect of romosozumab upon retreatment.

The OPTIMIST study is a two-year, randomised, active controlled, open-label, intervention trial. The study includes 270 postmenopausal women who will be randomised to 3 groups. Group 1 (n=90) will receive romosozumab for 12 months followed by zoledronate for 12 months. Group 2 (n=90) will receive romosozumab for 6 months followed by zoledronate for 12 months and romosozumab for 6 months. Group 3 (n=90 ) will receive romosozumab for 6 months followed by zoledronate for 18 months.

The investigational drugs in this study are romosozumab 210 mg/2,34 mL and zoledronate 5 mg/100 mL

This study will include 270 treatment naïve postmenopausal women. When inclusion and exclusion criteria have been reviewed, and the participant meets the requirements for study participation and continues to participate in the study, the patients will be randomized 1:1:1 Data will be registered in RedCAP (eCRF) and site monitoring assessed by the local Good Clinical Practice unit (GCP-unit).

The patients will be recruited from the outpatient clinics and the Dual-Energy X-ray Absorptiometry (DXA) units to which patients are referred from their general practitioner or fracture liaison services (FLS) at:

Department of Endocrinology, Odense University Hospital Department of Endocrinology and Internal Medicine, Aarhus University Hospital Department of Endocrinology, Køge Hospital Department of Endocrinology, Hvidovre Hospital Department of Endocrinology, Bispebjerg Hospital

During the intervention phase, there will be obtained fasting blood test, high-resolution peripheral quantitative computed tomography (HR-pQCT),Oral Glucose Tolerance Test (OGTT), DXA, Vertebral fracture assessment (VFA) and biochemistry at different time stamps. From 105 patients there will be obtained bone marrow aspirates and performed jamshidi bone biopsies.

The study will therefore show if it would be possible to treat twice as many patients for the same prize but also if the treatment for 12 months can be optimized. The knowledge about the optimal use of romosozumab will be included in an update of osteoporosis treatment guidelines. This will lead to optimized treatment of patients with severe osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (postmenopausal for at least two years)
* BMD T-score < -2.5 at lumbar spine, total hip, or femoral neck
* Osteoporotic fracture within the last 3 years at the spine, hip, pelvis, humerus or forearm after the age of 50 years.

Exclusion Criteria:

* Osteoporosis treatment including hormone replacement therapy within the last 5 years
* Metabolic bone disease
* Known disorders affecting bone metabolism, e.g., uncontrolled thyrotoxicosis, liver dysfunction (baseline phosphatase higher than twice upper limit), rheumatism, severe COPD (chronic obstructive pulmonary disease), hypopituitarism, Cushing's disease
* Ongoing treatment with glucocorticoids (systemic)
* Estimated glomerular filtration rate (eGFR) < 35 mL/min
* Contraindications for zoledronate according to the Supplementary protection certificates (SPC)
* Contraindications for romosozumab according to the SPC
* For the subgroup with Jamshidi biopsies contraindications for local anaesthetics according to the SPC
* For the subgroup with Jamshidi biopsies contraindications for tetracycline or doxycykline according to the SPC

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in total hip BMD | 24 months
  Change in total hip BMD

SECONDARY OUTCOMES:
Changes in femoral neck BMD | 24 months
  Change in femoral neck BMD
Changes in trabecular bone volume fraction (bone volume/tissue volume, BV/TV) and cortical porosity measured by high-resolution peripheral quantitative computed tomography (HR-pQCT) | 24 months
  Mean percent change in trabecular bone volume fraction and cortical porosity measured by HR-pQCT at the radius and tibia
Change in spine BMD | 24 months
  Change in spine BMD

OTHER OUTCOMES:
Bone resorption and formation -Changes in P1NP (procollagen type I N-terminal propeptide) | 1, 3, 6, 12, 18, 19, 21 and 24 months
  Changes in P1NP (blood sample)
Bone resorption and formation - Changes in CTX | 1, 3, 6, 12, 18, 19, 21 and 24 months
  Changes in cross-linked C-terminal telopeptide (CTX) (blood sample)
Bone resorption and formation - Changes in collagen | 1, 3, 6, 12, 18, 19, 21 and 24 months
  Bone turnover marker (BTM) collagen (blood sample)
Bone remodelling and modelling assessed using bone histology (jamshidi biopsy) | Month 1, 6, 18, 19, 24
  Investigate the activation of bone remodelling and modelling-based bone formation by ROMO assessed by bone histology (jamshidi biopsy) at 1 (any group), 6 (any group), 18 (group 3), 19 (group 2) and 24 (group 2) months. Biopsies will be obtained from 15 participants at each timepoint. Investigate the depletion of osteoprogenitor cells during ROMO treatment assessed by molecular bone histology and single-nucleic transcriptomics.
Investigate the number and composition of osteoprogenitor cells in the bone marrow during the first and second romosozumab treatment. | Month 1 and 19
  Investigate the number and composition of osteoprogenitor cells in the bone marrow during the first and second romosozumab treatment. Bone marrow (BM) aspirates will be obtained by aspiration of the iliac crest (10-15 ml) during the jamshidi biopsy.
Effect of romosozumab on glucose metabolism and insulin sensitivity (measurement of fasting glucose) | Month 1 and 3
  Change in fasting glucose (mmol/l) Blood sample
Effect of romosozumab on glucose metabolism and insulin sensitivity (measurement of Hba1c) | Month 1 and 3
  Change in glycated haemoglobin (Hba1c) (mmol/mol) Blood sample
Effect of romosozumab on glucose metabolism and insulin sensitivity (ogtt) | Month 1 and 3
  Change in oral Glucose tolerance test (OGTT) Data is collected by giving glucose and blood samples are taken afterward to determine the patients blood sugar (mmol/l) how quickly it is cleared from the blood
Effect of romosozumab on glucose metabolism and insulin sensitivity (HOMA-IR) | Month 1 and 3
  Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) calculated from fasting blood sugar (blood sample) and insulin levels (blood sample) by following equation: ([insulin (μU/ml)] × [fasting glucose (mmol/l)]/22,5)

CONTACTS AND LOCATIONS:
Overall Officials: Bente Langdahl, MD, Professor, DMSc, PhD,, Study Director — Department of Endocrinology and Internal medicin, Aarhus University Hospital
Locations (1):
- Department of Endrocinology and Internal Medicine, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No